CLINICAL TRIAL: NCT01289795
Title: Endothelial Function and Progenitor Cells in Acute Ischemic Stroke
Acronym: EPCAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Matthias Endres, MD, Center for Stroke Research Berlin
Other Study IDs: FF_NCRC_EPC01; 2009-010356-97 (EudraCT Number)
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-01

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases
MeSH Terms: conditions — Ischemic Stroke; Stroke; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, PBMC, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- first-ever ischemic stroke: first-ever ischemic stroke according to the WHO definition

SUMMARY:
The purpose of this study is to determine whether levels of circulating endothelial progenitor cells (cEPC) are increased in the acute phase of ischemic stroke.

DETAILED DESCRIPTION:
Endothelial dysfunction is a key component of atherosclerosis which contributes to the development of cardio- and cerebrovascular diseases. However, endothelial dysfunction (ED) is not established as a risk factor for ischemic stroke.

As a novelty the proposed trial investigates the following variety of indirect markers of endothelial function in acute ischemic stroke:

circulating endothelial progenitor cells (EPC), endothelial microparticles (EMP), ENDOPAT (RH- PAT ratio) in two regards:

1. time after ischemic events (< 48h, Days 4-5, day 7 or at discharge)
2. etiological stroke subtypes

It is not known whether these parameters are changed after acute cerebral ischemia and could possibly serve as specific target for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first ever ischemic stroke
* TIA, or transient symptoms with infarction (TSI)
* Age > or = 18 years old within 24 hours after onset
* Written informed consent to participate
* No evidence for dysphagia

Exclusion Criteria:

* Malignant hematopoietic disease (e.g. leukemia), severe systemic infections, severe immunological disease, renal or hepatic failure
* Pancreatitis, cholecystolithiasis, intestinal malabsorption
* Lactose intolerance
* Increased risk of aspiration
* Pregnancy
* Life expectancy less than 12 months
* Inability to give written informed consent
* Psychosis
* Alcohol dependency
* Abuse of illegal drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with first-ever ischemic stroke transferred to our stroke unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Levels of cEPC | <48h, day 4-5, discharge or day 7
  Levels of cEPC (CD34+/CD133+/VEGF2R+/CD31) in % of mononuclear cells using flow cytometry with respect to stroke subtypes.

SECONDARY OUTCOMES:
Levels of EMP | <48h, day 4-5, day 7 or discharge
  Levels of EMP (Annexin V+/CD31+; CD62E+) using flow cytometry with respect to stroke subtypes.
ENDOPAT | <48h, day 4-5,day 7
  Digital pulse volume change (with RH PAT as non invasive measurement (PAT-ratio; ENDOPAT, Itamar Medical Ltd.) for non-invasive, peripheral endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Endres, MD, Principal Investigator — Center for Stroke Research Berlin
Locations (1):
- Center for Stroke Research Berlin, Berlin, State of Berlin, Germany